

**Study Title:** An open-label, Phase 2 study to assess the safety and

efficacy of EQ101 in adult subjects with moderate to

severe alopecia areata

**Protocol Number:** EQ101-104-01

**Investigational Product(s):** EQ101

**Sponsor:** Equillium AUS Pty Ltd

**Development Phase:** Phase 2

NCT Number: NCT05589610

**Document Version Date:** 24 Apr 2024

## **CONFIDENTIAL**

Information contained in this protocol is proprietary and confidential in nature and may not be used, divulged, published, or otherwise disclosed to others except to the extent necessary to obtain approval of the Institutional Review Board/Independent Ethics Committee, or as required by law. Persons to whom this information is disclosed should be informed that this information is confidential and may not be further disclosed without the express permission of Equillium AUS Pty Ltd.



## STATISTICAL ANALYSIS PLAN

An open-label, Phase 2 study to assess the safety and efficacy of EQ101 in adult subjects with moderate to severe alopecia areata

**Protocol No.: EQ101-104-01** 





| 1 | TABLE OF CONTENTS | |
|---|---|---|
| 1 | Table of Contents | |
| 2 | List of Abbreviations | |
| 3 | Introduction | |
| 4 | | |
| | 4.1 Description of Study Design | |
| | 4.2 Objectives | |
| | 4.2.1 Primary Objectives and Endpoints | |
| | 4.2.2 Secondary Objectives and Endpoints | 7 |
| 6 | Statistical Considerations | |
| | 6.1 Standard Operating Procedures and Software | |
| | 6.2 General Considerations | 10 |
| | 6.3 Key Definitions | |
| | 6.4 Multiple Comparisons and Multiplicity | 11 |
| 7 | Analysis Populations | 16 |
| | 7.1 All Screened Population (ASP) | 16 |
| | 7.2 Safety Population (SP) | 16 |
| | 7.3 PK Analysis Population (PKAP) | 16 |
| 8 | Subject Screening, Enrolment and Disposition | 17 |
| 9 | Analysis population | |
| 11 | Demographics and Baseline characteristics | 20 |
| | 11.1 Demographics | 20 |
| | 11.2 Pregnancy and Follicle Stimulating Hormone (FSH) Test | 20 |
| | 11.3 Serology | |
| | 11.4 COVID-19 Test | |
| 12 | Medical History | 21 |
| 13 | Disease history | 22 |
| | Prior and Concomitant Medication | |
| 14 | | |
| 14<br>15 | Treatment Compliance and Exposure | 24 |
| | Efficacy | |
| 15 | Efficacy | 25 |
| 15<br>16 | 1 | 25<br>27 |
| 15<br>16 | Efficacy | 25<br>27 |
| 15<br>16 | Efficacy | 25<br>27<br>27 |
| 15<br>16 | Efficacy | 25<br>27<br>27<br>28 |
| 15<br>16 | Efficacy | 25<br>27<br>28<br>28<br>29 |
| 15<br>16 | Efficacy | 25<br>27<br>28<br>28<br>29 |
| 15<br>16<br>17 | Safety | 25<br>27<br>28<br>28<br>29 |

## LIST OF ABBREVIATIONS

| AA alopecia areata |
|---------------------------------------|
| alopecia areata |
| Anti-Drug Antibody |
| Adverse Event |
| Albumin |
| Alanine aminotransferase |
| Activated partial thromboplastin time |
| All Screened Population |
| Aspartate aminotransferase |
| Alopecia totalis |
| Anatomical Therapeutic Chemical |
| alopecia universalis |
| Body Mass Index |
| Calcium |
| Celiac Disease |
| Chloride |
| Clinician-Reported outcome |
| Coronavirus disease 2019 |
| Case Report Form |
| Clinically Significant |
| Clinical Study Report |
| coefficient of variation |
| Diastolic blood pressure |
| electronic data capture |
| Eyebrow |
| electrocardiogram |
| electronic Case Report Forms |
| Eyelash |
| End of study |
| End of Treatment |
| Follicle Stimulating Hormone |
| Good Clinical Practice |
| Hepatitis B core antibody |
| Hepatitis B surface antigen |
| hepatitis C virus |
| human immunodeficiency virus |
| International normalised ratio |
| immunophenotyping |
| Potassium |
| Mean corpuscular volume |
| Sodium |
| Neutralizing Anti-drug antibodies |
| Not Clinically Significant |
| polymerase chain reaction |
| pharmacodynamic |
| Pharmacodynamic Population |

| PK | pharmacokinetics |
|---------------------------|-------------------------------------------|
| PKAP | Pharmacokinetic Analysis Population |
| PoC | Proof of Concept |
| PRO | Patient-reported outcome |
| PT | Preferred Term |
| PTT Prothrombin time | |
| QTc Corrected QT interval | |
| QTcF | QTc using Fridericia's method |
| RAT | rapid antigen test |
| RBC | Red blood cell |
| SAEs | Serious Adverse Events |
| SALT | Severity of Alopecia Tool |
| SALT50 | 50% improvement of SALT |
| SALT75 | 75% improvement of SALT |
| SAP | Statistical Analysis Plan |
| SBP | Systolic blood pressure |
| SD | standard deviation |
| SOC | System Organ Class |
| SOPs | Standard Operating Procedures |
| SP | Safety Population |
| TB | tuberculosis |
| TEAEs | treatment-emergent adverse events |
| UN | Unknown |
| WBC | White blood cell |
| WHO-DD | World Health Organization Drug Dictionary |
| WOCBP | women of child-bearing potential |

## 3 INTRODUCTION

This Statistical Analysis Plan (SAP) provides the outline for the statistical analysis of the data collected for EQ101-104-01 protocol titled: "An open-label, Phase 2 study to assess the safety and efficacy of EQ101 in adult subjects with moderate to severe alopecia areata"

The SAP will be finalized prior to database lock. Any deviations from the SAP after database lock, reasons for such deviations, and all alternatives or additional statistical analyses that may be performed will be described in the Clinical Study Report (CSR).

#### 4 PROJECT OVERVIEW

#### 4.1 Description of Study Design

This is a multicenter, Phase 2, open-label Proof of Concept (PoC) study of EQ101 in adult subjects with at least 35% scalp hair loss due to alopecia areata (AA). Approximately 30 subjects will be enrolled in the study. During the 24-week treatment period, subjects will be dosed once weekly with EQ101 2 mg/kg Intravenous. Subjects will then be followed up for an additional 4 weeks after treatment. Randomisation and blinding have not been conducted in this study as this is a single-arm open-label PoC study.

### 4.2 Objectives

#### 4.2.1 Primary Objectives and Endpoints

The primary objective of this study is:

The primary objective of the study is to evaluate the safety and tolerability of EQ101 in adult subjects with moderate to severe AA over a 24-week treatment period.

The primary endpoints of this study are:

- Incidence, severity, and relationship of TEAEs, SAEs, TEAEs leading to discontinuation of study treatment.
- Changes in vital sign measurements
- · Changes in ECG parameters; and
- Changes in clinical laboratory results.

#### 4.2.2 Secondary Objectives and Endpoints

The secondary objectives of the study are:

- to evaluate the efficacy of EQ101 in adult subjects with moderate to severe AA over a 24week treatment period.
- to characterise the PK of EQ101 in adult subjects with moderate to severe AA.

#### 4.2.2.1 Efficacy

The primary efficacy endpoint is:

- The percent change from Baseline in Severity of Alopecia Tool (SALT) score at Week 24
   The secondary efficacy endpoints are:
- percent change from Baseline in SALT score at Weeks 4, 8, 12, 16, and 20.
- change from Baseline in SALT score at Weeks 4, 8, 12, 16, 20, and 24.
- percentages of subjects with a SALT ≤ 20 and those with a SALT ≤ 10 at Weeks 4, 8, 12, 16, 20, and 24.

- percentages of subjects achieving 30% (SALT<sub>30</sub>), 50% (SALT<sub>50</sub>), 75% (SALT<sub>75</sub>) and 90% (SALT<sub>90</sub>) improvement of SALT from Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- times to SALT score improvement of 30% (SALT<sub>30</sub>), 50% (SALT<sub>50</sub>) 75% (SALT<sub>75</sub>) and 90% (SALT<sub>90</sub>) improvement of SALT from Baseline.
- percentage of subjects achieving ClinRO Measure for eyebrow (EB) Hair Loss 0 or 1 with
   ≥ 2-point improvement from Baseline among subjects with ClinRO Measure for EB Hair
   Loss ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving ClinRO Measure for eyelash (EL) Hair Loss 0 or 1 with
   ≥ 2-point improvement from Baseline among subjects with ClinRO Measure for EL Hair
   Loss ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving ClinRO Measure for Body Hair Loss 0 or 1 with ≥ 2point improvement from Baseline among subjects with ClinRO Measure for Body Hair
  Loss ≥2 at Baseline and Week 24.
- percentage of subjects with Scalp Hair Assessment PRO of 0 or 1 with a ≥ 2-point improvement from Baseline among subjects with a score of ≥ 3 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving PRO measure for EB 0 or 1 with ≥ 2-point improvement from Baseline among subjects with PRO measure for EB ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving PRO measure for EL 0 or 1 with ≥2-point improvement from Baseline among subjects with PRO measure EL ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving PRO measure for Body Hair 0 or 1 with ≥ 2-point improvement from Baseline among subjects with PRO measure Body Hair ≥ 2 at Baseline and Week 24.

#### 4.2.2.2 Pharmacokinetics Endpoints

PK endpoints to be evaluated include (but are not limited to):

| • | plasma concentrations of EQ101 | and |
|---|--------------------------------------|----------|
| • | incidence of antidrug antibody (ADA) | |
| • | | <u> </u> |
| • | | |
| • | | |



#### 6 STATISTICAL CONSIDERATIONS

#### 6.1 Standard Operating Procedures and Software

Data will be handled and processed per the sponsor representative's Standard Operating Procedures (SOPs), which are written based on the principles of Good Clinical Practice (GCP).

All data conversions and statistical analyses will be performed using SAS® Version 9.4 or higher (SAS Institute, Cary, North Carolina, USA) with program code prepared specifically for the study by qualified Avance statisticians and SAS® programmers.

### 6.2 General Considerations

All data collected during the study (data originating from the electronic Case Report Forms (eCRFs) or electronic transfers will be presented in the data listings. Event-based listings will be sorted by subject identifier and event start date/time (i.e., Adverse Event (AE) start date/time). Assessment-based listings will be sorted by parameter name (alphabetically unless specifically stated otherwise), subject identifier, visit, assessment date and time (if applicable).

Unless otherwise stated, the following methods will be applied:

 <u>Continuous variables</u>: Descriptive statistics will include the number of non-missing values (n), arithmetic mean, standard deviation, median, minimum, and maximum values.

The minimum and maximum values will be displayed to the same decimal precision as the source data, the arithmetic mean and median values will be displayed to one more decimal than the source data, and the standard deviation (SD) values will be displayed to two more decimals than the source data for the specific variable.

The appropriate precision for derived variables will be determined based on the precision of the data on which the derivations are based, and statistics will be presented in accordance with the abovementioned rules.

- <u>Categorical variables</u>: Descriptive statistics will include frequencies and percentages
  per category. The denominator in all percentage calculations will be the number of
  subjects in the relevant analysis population, unless specifically stated otherwise.
  Percentages will be rounded to one decimal place and will not be displayed for zero
  frequencies.
- Repeat/unscheduled assessments: When values collected at scheduled study visits/time points is missing, repeat or unscheduled assessments closest to the scheduled visit date within the visit window defined in Table 1 and Table 2 will be used for the visit to calculate summary statistics in summary tables with visits as defined in section 6.6. All collected data will be included in the data listings. If an unscheduled visit was intended to replace the missing assessment for a scheduled visit this should be documented clearly before values are used as a scheduled visit assessment.
- <u>Assessment windows:</u> All assessments will be included in the data listings including
  additional safety labs collected and the protocol specified visit windows will not be
  applied to exclude assessments that were not performed on the protocol specified visit
  days. Visit information in the CRF will be used in the tables, listings, and figures.
- <u>Result display convention:</u> Results will be centre aligned in all summary tables and listings, subject numbers, visit, and parameter labels and comments may be left aligned

Protocol Number: EQ101-104-01 Document Status: Version 2.0

Version date: 24-Apr-2024

- Conversion of categorical values: In some instances, results may be with less than or greater than signs (i.e., < 9). The original source data captured will be displayed in the data listings (i.e., <9), while values may be converted to numbers which are half of the threshold value for summary table purposes. As an example, a value of < 9 may be converted to 4.5 before calculating summary statistics. In listings, the original value (i.e., < 9) is displayed instead of imputed values.
- Date and time display conventions: The following display conventions will be applied in all outputs where dates and/or times are displayed:

o Date only: YYYY-MM-DD

o Date and time: YYYY-MM-DD/HH:MM

If only partial information is available, unknown components of the date or time will be presented as UN (Unknown), for example "2022-UN-UN" or "UN:UN" for time.

#### 6.3 **Key Definitions**

The following definitions will be used:

- Date of the First Study Treatment Administration: The date of the first study treatment administration is defined as the earliest date on which a study treatment was administered.
- Baseline: The Baseline value is defined as the last available valid, non-missing observation for each subject prior to first study treatment administration on Day 1. If day 1 assessment has time missing, it will be considered as the baseline.
- Change from Baseline: The change from Baseline value at each visit will be calculated for all continuous parameters using the following formula when both values are available:

Change from Baseline Value = Result at specified visit – Baseline Value

% Change from Baseline: The % change from baseline value is defined as Change from Baseline divided by Baseline value. Study Day: The study day of an event is defined as the relative day of the event starting with the date of the first study treatment administration (reference date) as Day 1 (there will be no Day 0).

The study day of events occurring before the first study treatment administration will be calculated as:

Study Day = (Date of Event - Date of First Study Treatment Administration)

For events occurring on or after Day 1, study day will be calculated as:

Study Day = (Date of Event - Date of First Study Treatment Administration) + 1

Study days will only be calculated for events with complete dates and will be undefined for events that are 'Ongoing' at the end of the study.

#### 6.4 **Multiple Comparisons and Multiplicity**

No multiplicity adjustment will be carried out for this study.



#### **Adverse Events:**

For adverse events with unknown intensity (severity) or unknown relationship to study treatment, these will be imputed as follows:

- If the intensity (severity) of an adverse event is unknown/missing, the intensity will be imputed for the summary of adverse events as being the highest intensity, i.e., "Severe".
- If the relationship to investigational product of an adverse event is unknown/missing, the relationship will be imputed for the summary of adverse events as being "Related".

For adverse events, where either the onset time or end time (resolution time) is unknown, AE duration (in days) will be imputed as follows:

· If onset date is unknown

and it cannot be confirmed that onset was prior to the start of dose administration, then
the AE will be classified as treatment-emergent adverse events (TEAE), and AE
duration will be shown on the listing as UNKNOWN.

### • If onset time is unknown:

 If the date of onset is known to be same as the date of first dose administration, and it cannot be confirmed that onset was prior to the start of dose administration the AE will be reported as TEAE.



#### 6.6 Visit Display Conventions

## Visit Label for Summary Tables:

The following visit labels will be used in table summary outputs as applicable. Visit window defined in section 6.7 will be applied. :

- Screening
- Baseline
- Day 1 Post-dose
- ➤ Week 1
- ➤ Week 2
- ➤ Week 3
- ➤ Week 4
- ➤ Week 5
- ➤ Week 6
- ➤ Week 7
- ➤ Week 8
- ➤ Week 9
- ➤ Week 10
- ➤ Week 11
- ➤ Week 12
- ➤ Week 13
- ➤ Week 14
- ➤ Week 15
- ➤ Week 16
- ➤ Week 17
- ➤ Week 18
- ➤ Week 19
- ➤ Week 20
- ➤ Week 21
- ➤ Week 22.

➤ Week 23 ➤ Week 24 ➤ EOT¹ ➤ Week 28  $\triangleright$  EOS<sup>2</sup> Visit Label for Data Listings: For listings, CRF labels will be used.



## 7.1 All Screened Population (ASP)

Consists of all subjects who provided informed consent for the study.

## 7.2 Safety Population (SP)

Consists of all subjects who receive at least one dose of study drug. This analysis population is used for safety and efficacy analysis.

## 7.3 PK Analysis Population (PKAP)

Subjects in the safety population who have at least one measurable post-EQ101 exposure concentration.

## 8 SUBJECT SCREENING, ENROLMENT AND DISPOSITION

Subject enrolment information to be reported are listed below:

- Date of informed consent/reconsent
- Reconsent Version and Date
- Protocol Version
- Date of Eligibility Check at screening
- Subject ID

Subject disposition information to be reported are listed below:

- Subject ID
- Date received first study drug.
- Date of last Dose
- Study Completion Status
- Treatment Completion Status
- Date of Completion/ Discontinuation
- Reason for Discontinuation
- Date and reason for consent withdrawal

Counts and percentages for the number of Subjects Enrolled and Screen failed will be provided for the All Screened Population. Counts and percentages for the number of subjects dosed, Completed, withdrawn/Not Completed (with all reasons for not completion) treatment and study will be provided for the Safety Population.

Listings will be provided for the subject enrolment information (listed in above) and sorted by Subject ID for the All Screened Population. For the subject disposition information (listed in above), listings will be provided sorted by Subject ID for the Safety population, along with age, sex, race, and baseline weight (or Screening Weight for Screening Failures) of the Subject.

## 9 ANALYSIS POPULATION

The following analysis set information will be reported:

- Subjects included in Safety Population
- Subjects included in Pharmacokinetic Population



Counts and percentages for these Subjects under different analysis sets will be provided using the Safety Population

Listings of analysis population will be provided sorted by Subject ID for the Safety Population, along with age, sex, race, and baseline weight of the Subject.



#### 11 DEMOGRAPHICS AND BASELINE CHARACTERISTICS

#### 11.1 Demographics

The demographics variables to be reported are listed below:

- Age (years)
- Sex
- Women of child-bearing potential
- Race
- Ethnicity
- Weight (kg) at Screening
- Height (cm) at Screening
- Body Mass Index (BMI) (kg/m²) at Screening

Above variables will be summarized using descriptive statistics (specified in section 6.2) for Safety Population. Demographics variables will also be listed under Safety Population, sorted by Subject ID along with age, sex, race and baseline weight of the Subject.

## 11.2 Pregnancy and Follicle Stimulating Hormone (FSH) Test

All available pregnancy (serum or urine) and FSH test results will be displayed in data listing and sorted by Subject ID for Safety Population, along with age, sex, race, and baseline weight of the Subject.

#### 11.3 Serology

All available serology results (including human immunodeficiency virus (HIV), Hepatitis B surface antigen (HbsAg), Anti-hepatitis C virus (HCV) antibodies (if positive, HCV RNA measurement) will be displayed in data listing sorted by Subject ID for Safety Population, along with age, sex, race, and baseline weight of the Subject.

#### 11.4 COVID-19 Test

All available COVID-19 polymerase chain reaction (PCR) or rapid antigen test (RAT) test results will be displayed in data listing sorted by Subject ID for Safety Population, along with age, sex, race, and baseline weight of the Subject.

### 12 MEDICAL HISTORY

Medical history listings will be provided, sorted by Subject ID for Safety Population, along with age, sex, race, and baseline weight of the Subject. Medical history is coded using MedDRA 25.1.

The summary of medical history and medical history for subjects with autoimmune or mental health conditions will be presented by SOC in the order of descending frequency and PT within SOC in the order of descending frequency of the total column. Preferred term will be ordered by the total % and if they are tied, they are ordered alphabetically. The count and percentages of subjects with autoimmune disease or mental health conditions at End of Treatment/Early Termination compared to Screening will be summarised by SOC and PT for stable, improved or worsened. A Subject will only be counted once under a SOC or PT term by the worst status among multiple occurrences ("Worsened" is worse than "Stable" and "Stable" is worse than "Improved").

#### 13 DISEASE HISTORY

Disease history listings will be provided, sorted by Subject ID for Safety Population, along with age, sex, race, and baseline weight of the Subject. The summary of disease history will be presented by visit and following assessments for Safety Population.

The disease history information collected are as follows.

- Screening
  - Between 35% and 50% scalp hair loss, as determined by the Severity Alopecia Tool (SALT)
  - Alopecia Totalis
  - Alopecia Universalis
- Week 0, Day 1
  - Current AA Episode
    - What is the current Scalp involvement of the current AA episode (please specify the type)?
    - O Duration (<6 months, 6 months -1 year, >1 year -4 years and >4-7 years)
    - O Does the current AA episode affect the scalp only?
- Body Parts Affected by AA
  - o Eyelashes?
  - o If yes, duration
  - o Eyebrows?
  - o If yes, duration
  - o Body Hair (armpits, pubic hair, beard)?
  - o If Yes, please specify the area(s)
  - o If yes, duration
- Nail Changes
  - o Is subject experiencing nail changes currently?
  - o If yes:
    - Pitting
    - Koilonychia
    - Trachyonychia
    - Other
  - o If Yes, please specify the Duration for the most prominent/severe nail change

In addition, baseline SALT score and baseline SALT score categories of <50, >=50 to <95, and >=95 will be summarized using descriptive statistics.

Count and percentage of Alopecia Areata History Status at End of Treatment for nail disease and body hair disease will also be presented by stable, improved and worsened.

### 14 PRIOR AND CONCOMITANT MEDICATION

All medications will be coded by Anatomical Therapeutic Chemical (ATC) using World Health Organization Drug Dictionary (WHO-DD) (the version of WHODRUG GLOBAL B3 September 2022). The version used for coding will be specified in the footnote of the relevant outputs.

Prior medications are defined as those started before the start date/time of first study drug administration. Concomitant medications are defined as the medications taken at least once after the start date/time of first study drug administration, up to the end of study visit. If a clear determination cannot be made as to whether the medication is concomitant or not due to missing or incomplete data, the medication will be treated as concomitant medication taken during the study. Alopecia Areata Treatment History at Day 1 is also collected.

The number and percentage of Subjects using at least one concomitant medication will be displayed together with the number and percentage of Subjects using at least one medication within each anatomical therapeutic class (ATC-Level 1) and preferred name. It will be repeated for prior medication. Also the number and percentage of subjects with Alopecia Areata Treatment History at Day 1 will be summarized. These will be summarized under the Safety Population.

Listing of full details of prior and concomitant medications (medication taken, therapeutic class, Drug name, start and stop dates and times with ongoing status, indication, routes, frequency, dosage and due to AE) and concomitant procedure (procedure names, indication, and date of procedure) will be provided sorted by Subject ID for Safety Population, along with age, sex, race and baseline weight of the Subject, separately. Similarly, listing of full details of Alopecia Areata Treatment History at Day 1 will also be provided.

#### 15 TREATMENT COMPLIANCE AND EXPOSURE

All data collected in study drug administration eCRF will be included in the data listing. Listing of full details of treatment compliance and exposure (whether the subjects administered IP, Arm administered, Date and Time of administration, calculated dose, injection volume (mL), whether study drug administered per protocol and reason if no) will be provided sorted by Subject ID for Safety Population, along with age, sex, race, and baseline weight of the Subject.

Summary of Study Drug Administration will be provided for Safety Population. In the summary table, the summary statistics of total number of infusions, treatment duration (weeks), treatment duration (weeks) categories will be presented. Reasons for not dosing per protocol will be presented by visit (counts and percentages).

Treatment Duration (weeks) is calculated as (the last date of IP administration minus the first date of IP administration plus 7) divided by 7.

Treatment compliance (%) is defined as the number of infusions subject received\*100/24. Treatment compliance (%) will be presented descriptively. The number and percentage of subjects in each compliance category (0 - < 50 (%), 50 - <80 (%), 80 - <=100 (%)) will also be presented.

### 16 EFFICACY

Efficacy endpoints listed in 4.2.2.1 will be listed and summarised using the Safety Population. Summary statistics of change from baseline and percentage change from baseline for SALT Score will be presented.

Percentage and 95% confidence interval will be presented for the following efficacy endpoints.

- percentages of subjects with a SALT ≤ 20 and those with a SALT ≤ 10 at Weeks 4, 8, 12, 16, 20, and 24.
- percentages of subjects achieving 30% (SALT<sub>30</sub>), 50% (SALT<sub>50</sub>), 75% (SALT<sub>75</sub>) and 90% (SALT<sub>90</sub>) improvement of SALT from Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- times to SALT score improvement of 30% (SALT<sub>30</sub>), 50% (SALT<sub>50</sub>) 75% (SALT<sub>75</sub>) and 90% (SALT<sub>90</sub>) improvement of SALT from Baseline.
- percentage of subjects achieving ClinRO Measure for eyebrow (EB) Hair Loss 0 or 1\* with ≥ 2-point improvement from Baseline among subjects with ClinRO Measure for EB Hair Loss ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving ClinRO Measure for eyelash (EL) Hair Loss 0 or 1\* with ≥ 2-point improvement from Baseline among subjects with ClinRO Measure for EL Hair Loss ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving ClinRO Measure for Body Hair Loss 0 or 1\* with ≥ 2point improvement from Baseline at week 24 among subjects with ClinRO Measure for
  Body Hair Loss ≥2 at Baseline.
- percentage of subjects with Scalp Hair Assessment PRO of 0 or 1\* with a ≥ 2-point improvement from Baseline among subjects with a score of ≥ 3 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving PRO measure for EB 0 or 1\* with ≥ 2-point improvement from Baseline among subjects with PRO measure for EB ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving PRO measure for EL 0 or 1\* with ≥2-point improvement from Baseline among subjects with PRO measure EL ≥2 at Baseline at Weeks 4, 8, 12, 16, 20, and 24.
- percentage of subjects achieving PRO measure for Body Hair 0 or 1\* with ≥ 2-point improvement from Baseline at week 24 among subjects with PRO measure Body Hair ≥ 2 at Baseline.
- \* "0 point improvement from baseline", "1 point improvement from baseline", "≥2 points of improvement from baseline", and ""≥2 points of improvement from baseline with 0 or 1 point" will all be reported in summaries.

Time to SALT score improvement of 30% (SALT<sub>30</sub>), 50% (SALT<sub>50</sub>), 75% (SALT<sub>75</sub>), and 90% (SALT<sub>90</sub>) improvement will be summarised using the Kaplan-Meier method. For the subjects who did not achieve 30%, 50%, 75% or 90% SALT Score improvement, the week of the last SALT score assessment for the subject will be treated as censoring in these analyses. If there is no post-baseline assessment, the subject will be censored at date of first dose.

Subgroup analyses: SALT score, change from baseline and % change from baseline will be summarize by these subgroups:

- 1) By Demographics (age categories (<40, >=40), sex and race)
- 2) By Site
- 3) By Baseline SALT Score Categories (<50, >=50 < 95, >=95)
- 4) Duration of Current AA episode (<6 months, 6 months 1 year, > 1 year 4 years, >4 years 7 years)

SALT Score <=20 and <=10 and 30%, 50%, 75% and 90% improvement of SALT by visit will also be summarized by baseline SALT Score Categories (<50, >=50 - < 95, >=95).

A few SALT assessments were not assessed accurately (approval status of "No"). SALT assessments were reassessed for those cases. The SALT score analysis in this SAP is based on the SALT score data with approval status of "Yes".

For optional scalp biopsies, listing will be prepared sorted by subject identifier for the Safety population, along with age, sex, race, and baseline weight of the Subject.

For photographs for scalp, eyebrows and eyelashes and optional photographs of body hair (growth or regrowth) and fingernails, listing will be prepared sorted by subject identifier for the Safety population, along with age, sex, race, and baseline weight of the Subject.

#### 17 SAFETY

All safety endpoints will be analyzed using the Safety Population.

#### 17.1 Adverse Events

Adverse Events will be coded using the Medical Dictionary for Regulatory Activities MedDRA, Version 25.1. AEs that start during or after the first dose of study drug, or AEs with an onset prior to the first dose of study drug that worsen after study drug administration will be considered TEAEs.

Treatment-Related TEAEs are defined as any TEAEs reported with the causality of "Related" or missing to study treatment. All injection site reactions will be recorded as AE's and will be included in the AE tables and listings.

All AE summaries will be restricted to TEAEs only.

The TEAE summaries will include:

- Overall Summary of TEAEs
  - o TEAEs
  - Serious TEAEs
  - o TEAEs leading to study drug withdrawal
  - o TEAEs leading to study dose reduction
  - o TEAEs leading to study discontinuation
  - Any Serious TEAEs leading to Discontinuation from Study
  - Any Serious TEAEs leading to Death
  - o TEAEs by Severity (Grade 1 to Grade 5)
  - TEAE by Causality (Not related and Related)
  - Any Treatment-Related TEAEs
  - o Severity of Treatment-Related (Grade 1 to Grade 5)
- Summary by System Organ Class (SOC) and Preferred Term (PT)
  - o TEAEs
  - o TEAE summary for severity level (Grade 1 to Grade 5)
  - o TEAE by relationship with study drug (Unrelated versus Related)
  - Serious TEAEs
  - o Treatment-Related TEAEs
  - o Treatment-Related TEAEs for severity level (Grade 1 to Grade 5)
- Summary by PT
  - o TEAEs
  - Treatment-Related TEAEs



Version date: 24-Apr-2024

The above items will be presented using summary tables, which will include the number of events and the number of subjects (%) experiencing an event. If a subject experienced the same adverse event multiple times, this will only be counted once for the purpose of counting the number of subjects experiencing that adverse event.

Summary tables will be done for the Safety population. Where SOC and PT are reported, the display will be sorted by the descending order by total counts for SOC and then by PT. All AEs will be listed and will include the verbatim term, PT, SOC, treatment, causality/severity, date and time of consent, date and time of resolution, outcome, infusion site reaction, infusion related reaction and/or hypersensitivity reactions, action taken, discontinuation from study, SAE, TEAE, concomitant medications, additional treatment given, other action taken, worsening of medical history and the terms of the corresponding medical history, whether the adverse event associated with a congenital anomaly or birth defect, whether the adverse event result in persistent or significant disability or incapacity, whether the AE result in death, whether the adverse event result in initial or prolonged hospitalization for the patient, whether the AE was life threatening, and whether the adverse event associated with other serious or important medical events. Separate listings will be created for SAEs, Adverse Events Leading to Study Dose Reduction, Study Drug Withdrawal, and Discontinuation from study, and Infusion Site Reactions, infusion related reactions and/or hypersensitivity reactions. These listings will be presented by Subject ID and date for the Safety Population, along with age, sex, race, and baseline weight of the subject. Listing of death will be presented for the Safety Population if there was any death reported in the study.

#### 17.2 Safety Laboratory Assessments

For the haematology, serum chemistry and coagulation, continuous data summary statistics (as described in Section 6.2) and count and percentages of normal and abnormal (defined by a testspecific normal range) will be presented for values, change from baseline at each visit.

In addition, Shift from Baseline at each visit for haematology, serum chemistry and coagulation lab parameters (low, normal, high) will also be presented using counts and percentages in shift tables.

For urinalysis and urine microscopy, continuous data summary statistics (as described in Section 6.2) and count and percentages of normal and abnormal will be presented for values at each visit.

The listings of laboratory parameters (haematology, serum chemistry, coagulation, and urinalysis) will include all the information collected. In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values (where applicable) at each post baseline (scheduled and unscheduled) visit will be presented. These listings will be presented sorted by Subject ID and assessment date for the Safety Population, along with age, sex, race, and baseline weight of the subject.

#### 17.3 **Vital Sign Assessments**

The following vital signs measurements will be summarised at the time points specified in the study schedule of events (Section 24):

- Heart Rate (beats/mins)
- Systolic blood pressure (SBP) (mmHg)
- Diastolic blood pressure (DBP) (mmHg)

- Body Temperature (°C)
- Body Weight

Summary statistics for vital sign parameters in accordance with Section 6.2 will be presented for baseline and for each scheduled post-baseline visit (which also includes change from baseline). These summary tables will be done for Safety Population.

The listing of vital sign parameters will include all the information collected. In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values at each post baseline (scheduled and unscheduled) visit will be presented. This listing will be presented sorted by Subject ID and assessment date/time for the Safety Population, along with the age, race, and baseline weight of the subject.

## 17.4 12-Lead Electrocardiogram (ECG)

The following ECG measurements will be summarised at the time points specified in the study procedure schedule:

- Heart Rate (bpm)
- PR interval (msec)
- QT interval (msec)
- QRS interval (msec)
- QTcF interval (msec)
- Clinical Interpretation

Summary statistics for ECG parameters in accordance with Section 6.2 will be presented for baseline and for each scheduled post baseline visit (which also includes the change from baseline). In addition, clinical result (Normal, Abnormal not clinically significant, abnormal, and clinically significant) will be summarized by counts and percentages for baseline and for each scheduled post baseline visit. These summary tables will be done for Safety Population.

The listing of ECG parameters will include all the information collected. In addition, the observations that are used as the baseline record (value) for each parameter will be flagged, and the change from baseline values at each post baseline (scheduled and unscheduled) visit will be presented. This listing will be presented sorted by Subject ID and assessment date/time for the Safety Population, along with the with the age, race, and baseline weight of the subject.

### 17.5 Physical Examinations

The listing of physical examinations (including full and symptom directed examinations) will include all the information collected. This listing will be presented sorted by Subject ID and assessment date/time for the Safety Population, along with the age, race, and baseline weight of the subject.

## 18 PHARMACOKINETICS

Plasma concentrations of EQ101 will be provided after DBL. Concentration data can be reported outside the scope of this SAP as additional listings for individual subjects and as statistical summaries grouped by the scheduled timepoint and provided separately after the DBL. The statistical summary may include mean, standard deviation (SD), coefficient of variation (CV%), maximum, minimum, median, geometric mean, and geometric CV%.







# 23 FINAL ANALYSIS (END OF STUDY)

The final analysis will be conducted after all subjects have completed the study, the clinical database has been locked, and the analysis populations have been approved.

The final analysis will be based on the final version of the SAP. Any deviations from the planned analysis will be documented in the CSR.









